CLINICAL TRIAL: NCT04915469
Title: Evaluation of Enhanced Adherence Counseling as a Strategy to Optimize Adherence, Retention and Viral Suppression Among Children and Adolescents, in Homa Bay County, Kenya
Brief Title: Enhanced Adherence Counselling, Pre-Post Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rose Otieno Masaba, Associate Director Public Health Evaluations, Elizabeth Glaser Pediatric AIDS Foundation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EG0202
Record Dates: First submitted 2021-05-27; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: HIV Infection
Keywords: Children; Adolescents; Viral suppression; Antiretroviral therapy
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: This is a pre-post study design. The post-group receive an intervention of a standardized enhanced adherence counseling package
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-standardization group (No Intervention): Pre intervention- patient level data are abstracted retrospectively from the charts of patients with VL >1000 copies/ml on demographic characteristics and clinical outcomes and facility level data from summary forms for up to 24 months prior to the implementation of the standardized EAC package.
- Post-standardization group (Other): This group of participants will receive the standardized enhanced adherence package. After implementation of the standardized EAC package, data will be prospectively collected from participants with high viral load (>1000 copies).
  Interventions: Other: Standardized enhanced adherence counseling package

INTERVENTIONS:
Other: Standardized enhanced adherence counseling package — A standardized package was developed to support the adherence counsellor and other cadres to ensure provision of quality EAC sessions for children, adolescents and their caregivers. The package included; 1) Orientation and on job mentorship on EAC processes to clinicians, nurses, peer educators and mentor mothers. 2) Using a communication's training curriculum, providers were trained on psychosocial support and communication skills for children and their caregivers. 3) Appointment management was done using appointment dairies or a digital platform that sends patients short message services (SMS) reminders 3 days and 1 day before a scheduled clinic day. 4)Home visits. - All home visits were done according to the EGPAF standard operation procedures (SOPs) drawn from the Kenya National guidelines. 5) Individualized case management -Each EAC client was allocated a case manager who ensured that the barriers to adherence were identified and tackled both at individual and community level.
  Arms: Post-standardization group

SUMMARY:
Viral suppression among children and adolescents in Kenya is currently sub-optimal at 60% and 63% respectively. Under the current Kenya Ministry of Health Guidelines, clients with viral load of >1000 copies/ml, should receive a minimum of three enhanced adherence counselling (EAC) sessions offered every two weeks and have a repeat viral load conducted 3 months after EAC completion. However, delivery of the EAC is not standardized and there is limited data available to evaluate the effectiveness of the three counselling sessions. Observational data from Elizabeth Glaser Pediatric AIDS Foundation (EGPAF)-supported sites in Homa Bay and Turkana counties indicate that among children and adolescents with a viral load > 1000 copies/ml, approximately 40% received the recommended three minimum EAC sessions and, after receiving EAC sessions, viral suppression was 33% in children aged below 9 years, 27% in adolescents aged between 10-14 years, 38% in adolescents aged 15 to 19 years and 53% in adults. The investigators propose to evaluate the implementation, effectiveness and acceptability of a standardized EAC package implemented at EGPAF-supported sites.

Methods: The investigators will use mixed methods to evaluate specific clinical outcomes (viral suppression) adherence, retention) among children and adolescents who receive the EAC package after suspected treatment failure, and if applicable, after switch to second and third line. The investigators will use a pre/post intervention assessment to evaluate the effectiveness of the EAC package, and qualitative methods (in-depth individual interviews (IDI) and focus group discussions (FGD)) to identify facilitators and barriers to accessing EAC. A process evaluation will be conducted to determine whether the standardized EAC package has been implemented as intended across sites. The study population is defined as children aged 0-19 years receiving Antiretroviral therapy (ART) in selected EGPAF supported sites.

Policy Significance:

Dissemination of findings will be done through: internal evaluation report shared with stakeholders, donors, and the Ministry of Health (MOH) and abstracts presented at local and international conferences; and, manuscripts for publication in peer-reviewed journals. Findings are expected to inform the continuous review and improvement of HIV Program delivery in Kenya, as the ministry of health and partners strive to meet international standards.

DETAILED DESCRIPTION:
BACKGROUND Viral suppression is a proxy for successful anti-retroviral therapy (ART) and is the "3rd 90" of the (Joint United Nations Programme on HIV/AIDS (UNAIDS) 90-90-90 strategy. In Kenya, viral suppression among children and adolescents is sub-optimal at 60% and 63% respectively. Potential barriers to viral suppression can be individual (knowledge deficit, side effects, forgetting, substance abuse, depression, and pill burden), social (stigma, food insecurity, and family relationships) and structural (clinic frequency, school, relationship with health worker, long waiting times and lack of dose adjustment). Enhanced adherence counselling (EAC) aims to identify and address barriers to adherence to enable viral suppression. Following a client viral load of >1000 copies/ml, the Kenyan 2016 antiretroviral therapy guidelines recommend a minimum of three EAC sessions offered two weeks apart. Changes in viral load are detected through a repeat test conducted 3 months after EAC. Clients with repeat VL < 1000 are considered to be virally suppressed and are, therefore, maintained on the same Antiretroviral(ARV)drug regimen. Clients with persistent viral load above 1000 copies/ml are deemed to have failed first-line treatment, and are thereafter, switched to the appropriate second line or third line ARV drug regimen.

Delivery of the EAC is not standardized and there is limited data available to evaluate the effectiveness of the three counselling sessions. Observational data from EGPAF-supported sites in Homa Bay and Turkana counties indicates that for children and adolescents with a viral load > 1000 copies/ml, approximately only 40 percent received the recommended three minimum EAC sessions. Following EAC, viral suppression was 33% in children aged below 9 years, 27% in adolescents aged between 10-14 years, 38% in adolescents aged 15 to 19 years and 53% in adults. The investigators propose to evaluate the implementation, effectiveness and acceptability of a standardized EAC package implemented at EGPAF-supported sites in Homa Bay County.

Adherence to ART among Children with HIV in Kenya An estimated 98,000 children aged between 0-14 years are infected with HIV in Kenya. HIV/AIDS accounts for 15% of mortality among children less than 5 years of age, while 50-60% of children infected with HIV at birth die before their second birthday.

Adherence to ART, retention in care and achieving viral suppression are substantial challenges in the management of infants and children on ART. Infants and children rely on others to administer their medications and to ensure clinic attendance. Caregivers may face barriers that can reduce medication adherence and clinic attendance. Some caregivers place too much responsibility for managing medications on older children and adolescents before they are developmentally able to undertake such tasks. Adherence may also be jeopardized by social and health issues within a family (e.g. substance abuse, poor physical or mental health, unstable family relations, and poverty). To improve outcomes for infants and children on ART, Kenya guidelines recommend provision of caregiver education to all parents/guardians of children receiving ART. To this end, a caregiver-specific treatment literacy curriculum has been developed by the MOH for caregiver training.

Guidelines on use of Antiretroviral Drugs for Treating and Preventing HIV Infection in Kenya.

The 2016 Kenya Ministry of Health guidelines on the use of ART for treating and preventing HIV recommend that ART should be started in all patients as soon as possible, preferably within 2 weeks after confirmation of HIV infection. A patient preparedness assessment is completed prior to initiating ART. Adherence support mechanisms need to be put in place for same day ART initiation. Routine monitoring of treatment response in adults, adolescents and children older than 2 years includes as assessment of VL at 6 months after ART initiation and 12 months after initiation of ART, and if suppressed (VL<1000 copies/ml3), annually thereafter. Routine monitoring for infants, and children below 2 years is recommended at baseline, 6 months and 12 months after initiation of ART, then annually thereafter if the patient is stable and virally suppressed. Targeted VL is done for patients with suspected treatment failure. Targeted VL is also done when considering regimen change or single drug substitutions in patients who have been on ART for at least 6 months.

For patients with persistently high VL (>1,000 copies/ml) after 6 months after initiating ART, and for those who were previously suppressed but found to have high viral load (VL>1000 copies/ml) after more than 6 months after initiating ART, the guidelines recommend at least 3 patient-focused enhanced adherence counselling sessions within a 3-month period to address possible barriers before repeating the viral load test

Evaluation Goals and Objectives Goal: To evaluate clinical outcomes (viral suppression, adherence, retention) among children and adolescents with suspected treatment failure who receive the standardized enhanced adherence counselling package as compared to clinical outcomes for children and adolescents with suspected treatment failure who received services before standardization of enhanced adherence counselling package.

Overview of Evaluation Design This study uses a mixed method design. The investigators will use a pre-post design to evaluate specific treatment outcomes among children and adolescents receiving the standardized EAC package after suspected treatment failure and after switch to second- and third-line drug regimens. The investigators will conduct qualitative interviews and abstract patient outcome data to evaluate the effectiveness of the standardized EAC package, and qualitative methods (in-depth individual interviews and focus group discussions) to identify facilitators and barriers to accessing EAC. A process evaluation will be conducted to determine whether the standardized package of EAC was implemented as intended.

The study will use both qualitative and quantitative data collection and analysis methods. Pre-intervention, the investigators will abstract patient level data retrospectively from the charts of patients with VL >1000 copies/ml on demographic characteristics and clinical outcomes and facility level data from summary forms for up to 24 months prior to the implementation of the standardized EAC package. Viral suppression will be evaluated at 6 and 12 months. After implementation of the standardized EAC package, data will be prospectively collected from participants with high viral load (>1000 copies). After receiving the standardized EAC package, participants who are not suppressed will be switched to either second or third line and data will be collected prospectively from them at every visit. The investigators will use quantitative and qualitative methods of individual interviews, focus group discussions, and patient satisfaction surveys to assess acceptability of EAC and related services, as well as perceptions of facilitators and barriers to services pre and post intervention. Data related to EAC coverage will be abstracted from facility records. Coverage is defined as the proportion of patients with suspected treatment failure (STF) who receive a repeat viral load. A repeat viral load is only done after the completion of EAC and good adherence. Timelines will be determined using time from date when first high VL is documented in patient's chart to date of standardized EAC intervention (initiation and completion). This information will be abstracted from patient charts.

Study Population The study population will include HIV-positive male and female children and adolescents aged 0-19 years who are enrolled on ART at EGPAF supported sites and have suspected treatment failure. The investigators will interview parents/caregivers, peer educators/adherence counselors and health care providers in the same facilities to assess the barriers and facilitators, including satisfaction with care, to accessing EAC, both pre and post-intervention. For children below 9 years, the investigators will interview their caregivers.

. Sites Selection There are 171 facilities supported by EGPAF under the Timiza90 project in Homa Bay County. Among these, the investigators purposively selected seven high-volume facilities in order to provide sufficient numbers of children and adolescents with suspected treatment failure to include in the evaluation.

Sample size and Sampling Strategy The investigators purposively selected facilities that had the greatest number of unsuppressed patients based on viral load tests done between October 2017 to September 2018. In the selected facilities, the investigators captured data from the records of all patients who were unsuppressed over the period Oct 2016 - Sep 2018, (pre-intervention). Similarly, investigators captured data from the records of all patients who were unsuppressed for the post-implementation period, February 2019 - September 2020.

Sample size was calculated with an estimated 80% power at a 95% confidence level to demonstrate a minimum 10% increase in viral suppression due to the standardized EAC, adjusted for facility clustering (design effect 1.5), and estimates of missing records or lost to follow-up (+20%). The investigators used probability proportional-to-size sampling, based on the volume of VL tests by facility and age group; 0-9, 10-14, 15-19 years.

The investigators assume a 4:1 pre/post implementation number of clients unsuppressed for the 0-9-year age group and 3:1 pre/post implementation number of clients unsuppressed for the 10-14- and 15-19- year age groups. Table 3 presents these data, considering missing records for the retrospective cohort, or lost-to-follow up/missing records for prospective/post-intervention cohort, which may subsequently reduce the power to be able to demonstrate a difference. These estimates are unadjusted for facility clustering; the investigators will adjust for any clustering in the analysis.

Challenges and limitations Challenges and limitations to the evaluation include the quality of the patient records and their potential for missing data, the potential for response and response bias, the need for skilled interviewers and facilitators for the interviews and FGDs.

Analysis of patients' record data may be limited by poor data quality including missing data and data entry error especially for the retrospective data. The amount and patterns of missing data will be evaluated and appropriate statistical methods, as they may be applicable, will be used to account for the missing data in the analyses. The investigators will mitigate error resulting from data entry by re-entering a 5 percent random sample of the records on an ongoing basis. This subsequent data entry will be carried out by a different data entry clerk from the original clerk. Deviations of >10 percent will result in retraining of the data entry staff.

Challenges with FGDs and IDIs include the potential for response bias, (the respondents may report what the interview would like to hear), differential non-response, (participants who refuse to be interviewed may be different to those who agree), and recall bias, (participants may selectively recall stakeholders and events).

ELIGIBILITY:
Inclusion Criteria for children and adolescents

* Age 0-19 years
* HIV positive
* On ART for at least 6 months
* Last VL >1000 copies
* Parental/guardian consent
* Assent (for 10-17-year old)
* Consent (for 18-19-year old)

Inclusion criteria for parents/caregivers

* Parent/guardian to a child/adolescent on ART with VL>1000 copies
* Provides consent

Inclusion criteria for service providers, Peer educators, Adherence/Psychosocial support counselors

* Working in the facility for at least 3 months
* Provides services to HIV positive children and adolescents on ART
* Provides consent

Exclusion Criteria:

* Already receiving EAC
* Receiving services at non-participating facility
* Not providing HIV services to children and adolescent

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 741 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
Viral Suppression | This will be done after 3 months of EAC
  Viral load will be done following completion of at least 3 enhanced adherence counselling sessions. a patient with a viral load less than 1000 copies/ml3, will be considered to have suppressed

SECONDARY OUTCOMES:
Adherence to clinic visits and pharmacy pick-ups | 9 months
  A patient will be considered to have adhered to clinic visits and pharmacy pick-ups if they came to the clinic for their visits and medication pick-ups on the actual appointment date.
Retention on ART | At 9 months
  A patient is considered retained if s/he visited the facility within the last 90 days and actively on ART medication and not documented to have died or transferred out.
Lost to follow-up(LTFU) | At 9 months
  A patient will be considered LTFU if absent from the facility for more than 90 days after the last scheduled follow up date and there was no documentation of death or transfer out and 3 failed attempts to contact either by phone or physically
Time to 1st EAC following diagnosis of suspected treatment failure | baseline
  Diagnosis of suspected treatment failure is defined by the date the high viral load is documented in the patients' chart)
Average time to completion of EAC sessions | at 3 months
  Time taken to complete EAC sessions leading to either suppression or a switch of regimen

CONTACTS AND LOCATIONS:
Overall Officials: Rose Masaba, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation
Locations (1):
- Homa Bay county, Homa Bay, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gill MM, Ndimbii JN, Otieno-Masaba R, Ouma M, Jabuto S, Ochanda B. Adherence challenges and opportunities for optimizing care through enhanced adherence counseling for adolescents with suspected HIV treatment failure in Kenya. BMC Health Serv Res. 2022 Jul 29;22(1):962. doi: 10.1186/s12913-022-08373-9. PMID 35906574